CLINICAL TRIAL: NCT03633461
Title: Multicenter, Randomized, Controlled, Double-Masked Clinical Trial to Evaluate the Efficacy of OC-02 Nasal Spray on Signs and Symptoms of Dry Eye Disease (the RAINIER Study)
Brief Title: Evaluation of the Efficacy of OC-02 Nasal Spray on Signs and Symptoms of Dry Eye Disease (the RAINIER Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oyster Point Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPP-003
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Results first posted 2022-02-03 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OC-02 (simpinicline) spray spray, 11.1 mg/ml (Active Comparator): OC-02 (simpinicline) nasal spray, 11.1 mg/ml
  Interventions: Drug: OC-02 (simpinicline) nasal spray
- Placebo (Placebo Comparator): Placebo (vehicle) nasal spray
  Interventions: Drug: Placebo (vehicle) nasal spray

INTERVENTIONS:
Drug: OC-02 (simpinicline) nasal spray — OC-02 (simpinicline) nasal spray, 11.1 mg/ml
  Other Names: OC-02 (simpinicline) nasal spray, 11.1 mg/ml
  Arms: OC-02 (simpinicline) spray spray, 11.1 mg/ml
Drug: Placebo (vehicle) nasal spray — Placebo (vehicle) nasal spray
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of OC-02 nasal spray compared to placebo on signs and symptoms of dry eye disease (DED).

DETAILED DESCRIPTION:
This was a Phase 2, multicenter, randomized, double-masked, placebo-controlled study designed to evaluate the safety and efficacy of OC-02 Nasal Spray in adult subjects with dry eye disease. Approximately 45 subjects, at least 22 years of age, with a history of dry eye disease and meeting all other study eligibility criteria were planned to be randomized to receive an application of OC-02 or placebo twice daily (BID) for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have used and/or desired to use an artificial tear substitute for dry eye symptoms within 60 days prior to Visit 1

Exclusion Criteria:

* Have had any intraocular surgery (such as cataract surgery), extraocular surgery (such as blepharoplasty) in either eye within three months or refractive surgery (e.g. laser epithelial keratomileusis, laser-assisted in-situ keratomileusis, photorefractive keratectomy or corneal implant) within twelve months of Visit 1
* Have a history or presence of any ocular disorder or condition in either eye that would, in the opinion of the Investigator, likely interfere with the interpretation of the study results or participant safety such as significant corneal or conjunctival scarring; pterygium or nodular pinguecula; current ocular infection, conjunctivitis, or inflammation not associated with dry eye; anterior (epithelial) basement membrane corneal dystrophy or other clinically significant corneal dystrophy or degeneration; ocular herpetic infection; evidence of keratoconus; etc. Blepharitis not requiring treatment and mild meibomian gland disease that are typically associated with dry eye disease are allowed.
* Have a systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study or with the lengthier assessments required by the study (e.g., current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction or heart disease, etc.)
* Have a known hypersensitivity to any of the procedural agents or study drug components
* Have any condition or history that, in the opinion of the investigator, may interfere with study compliance, outcome measures, safety parameters, and/or the general medical condition of the subject

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Louisville, Louisville, Kentucky
  - Nashville, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OC-02 (Simpinicline) Spray Spray, 11.1 mg/ml | Placebo
Started | 34 | 19
Completed | 34 | 18
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Subjects in the ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | OC-02 (Simpinicline) Spray Spray, 11.1 mg/ml | Placebo | Total
Number analyzed (Participants) | 34 | 19 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (13.5) | 64.7 (11.5) | 63.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 15 | 42
  Male | 7 | 4 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black/African American | 4 | 0 | 4
  White | 29 | 19 | 48
  Not Hispanic/Latino | 31 | 18 | 49
  Hispanic/Latino | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 34 | 19 | 53
Schirmer's Test [Mean (Standard Deviation); unit: mm] — The Schirmer's test measures the amount of tears produced by placing a paper strip in the eye for 5 minutes and distance of wetting was recorded. Schirmer's test scores from 0-35 mm where a higher score is indicative of a better outcome.
  mm | 6.3 (3.1) | 5.1 (3.1) | 5.9 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Schirmer's Test From Baseline to 28 Days
Description: The primary end point was the change in anesthetized Schirmer's Test Score (STS) from baseline to 28 days in the study eye following treatment with OC-02. Schirmer's test score from 0-35 mm where a higher score is indicative of a better outcome.
Time Frame: 28 days [Visit 1 (baseline) and Visit 5 (28 Days)]
Population: Subjects in the ITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | OC-02 (Simpinicline) Spray Spray, 11.1 mg/ml | Placebo
Number analyzed (Participants) | 34 | 18
mm | 10.5 [7.4 to 13.5] | 5.7 [1.4 to 9.9]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the first dose of study drug administration until the final study visit at Visit 5 (28 days)
Arm/Group | OC-02 (Simpinicline) Spray Spray, 11.1 mg/ml | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/19
Other Adverse Events (participants affected / at risk) | 33/34 | 11/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OC-02 (Simpinicline) Spray Spray, 11.1 mg/ml (N=34) | Placebo (N=19)
Visual acuity reduced (Eye disorders) | 3 | 0
Vision blurred (Eye disorders) | 0 | 2
Eye irritation (Eye disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 22 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal inflamation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Instillation site irritation (General disorders) | 4 | 0
Instillation site paresthesia (General disorders) | 1 | 0
Aphtous ulcer (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 1
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 3 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT03633461/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT03633461/SAP_001.pdf